CLINICAL TRIAL: NCT05275517
Title: Investigation of the Relationships Between Physical Activity Level, Quality of Life and Cognitive Level in Breast Cancer Patients
Brief Title: The Relationships Between Physical Activity Level, Quality of Life and Cognitive Level in Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Nazan Ozturk, Principal Investigator, Aydin Adnan Menderes University
Other Study IDs: İboelif22
Record Dates: First submitted 2022-02-10; First posted 2022-03-11 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Physical Activity; Patient; Quality of Life; Chemotherapy
Keywords: Physical Activity; Quality of Life; Chemotherapy; Cognitive level
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to determine the relationships between physical activity level, quality of life and cognitive level in patients with breast cancer and to compare the results with a population of similar age group.

DETAILED DESCRIPTION:
This study is a cross-sectional, analytical type study and will be conducted with chemotherapy patients diagnosed with breast cancer and treated in Aydın Adnan Menderes University Faculty of Medicine Research and Practice Hospital, Department of Oncology. Patients diagnosed with breast cancer and undergoing chemotherapy will be provided by the researcher to fill out the questionnaires.

Healthy peers will also form the control group. First of all, mini mental test will be applied to all participants and those who get at least 24 points from the test will be included in the study. International Survey of Physical Activity (IPAQ),EORTC QLQC30 Quality of Life Scale,Montreal Cognitive Assessment Scale (MOCA) will be administered to all participants face to face by the researcher.

The hypotheses the investigators will test for this purpors; H0; There is no relationship between physical activity level, quality of life and cognitive level in patients with breast cancer.

H1a: Physical activity level of patients with breast cancer affects their quality of life.

H1b: Physical activity level affects cognitive level in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Being treated at Aydın Adnan Menderes University Faculty of Medicine Research and Application Hospital
* Being diagnosed with cancer at least 3 months before the study and receiving chemotherapy treatment
* Mini mental test result of at least 24
* To be conscious,
* Be over the age of 18,
* Being diagnosed with mass-style cancer,
* Patients with walking function

In the Healthy Control group:

* Over 18 years
* Never been diagnosed and treated for cancer before
* Volunteers who do not have a disease that will impair cognitive functions

Exclusion Criteria:

* Patients with brain metastases
* Patients with cognitive and psychiatric problems
* Patients with a diagnosis of hematological type cancer
* Patients receiving palliative care will not be included in the study. For the healthy control group
* With systemic disease
* Have a chronic illness
* Having problems that interfere with physical activity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients receiving chemotherapy with the diagnosis of breast cancer in the Oncology Department of Aydin Adnan Menderes University Research and Practice Hospital
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Demographic Information Form | 1 year
  In the form prepared by the researchers with the support of the literature, there are questions about the sociodemographic characteristics of the participants such as gender, age, height, weight, educational status,etc.
Mini Mental State Test | 1 year
  It is a scale used to evaluate the cognitive status of individuals. Test; It evaluates verbal responses including attention, orientation and memory, ability to obey verbal and written orders, write spontaneous sentences, and copy a complex drawing. The cut-off value of this scale, which consists of a total of 30 points, is 24 points. Values below 24 indicate deterioration in cognitive status.
International Survey of Physical Activity (IPAQ) | 1 year
  This form will be used to determine the duration of physical activity that patients have done in the last 7 days. The 27-question survey evaluates in detail the amount of walking done in the past week and the amount of moderate to vigorous physical activity done at work, transportation, housework, gardening and leisure activities.
EORTC QLQC30 Quality of Life Scale | 1 year
  This questionnaire is used to determine their quality of life. It includes 30 questions and three subheadings: general well-being, functional difficulties and symptom control. The first 28 of the 30 items in the scale are a four-point Likert-type scale and the items are evaluated as Never: 1, A little: 2, Quite: 3 or A lot: 4 points.
Montreal Cognitive Assessment Scale (MOCA) | 1 year
  This test assesses different cognitive functions including attention and concentration, executive functions, language, memory, visual construction skills, abstract thinking, calculation and orientation. The highest score that can be obtained from the test is 30. Cognitive status levels of individuals with a score of 21 and above are considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Nazan Ozturk, PhD., Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Aydın Adnan Menderes University Hospital, Aydin, Turkey (Türkiye)